CLINICAL TRIAL: NCT06719336
Title: Addition of High-dose Hyperfractionated Simultaneous Integrated Boost Radiotherapy to the Maintenance Therapy with PD-L1 Inhibitor Versus PD-L1 Inhibitor Alone for Extensive Stage Small Cell Lung Cancer (STONE-001)
Brief Title: Addition of Thoracic Consolidation Radiotherapy to the Maintenance Immunotherapy for ES-SCLC (STONE-001)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Shi, MD (Other)
Responsible Party: Sponsor-Investigator, Anhui Shi, MD, Chief Physician of Radiotherapy Department, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STONE-001
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: Extensive-stage small cell lung cancer; Thoracic consolidation radiotherapy; Immune Therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Addition of thoracic consolidation radiotherapy to the maintenance therapy with PD-L1 inhibitor (Experimental)
  Interventions: Radiation: High-dose Hyperfractionated Simultaneous Integrated Boost Radiotherapy; Drug: atezolizumab or durvalumab
- Maintenance therapy with PD-L1 inhibitor (Active Comparator)
  Interventions: Drug: atezolizumab or durvalumab

INTERVENTIONS:
Radiation: High-dose Hyperfractionated Simultaneous Integrated Boost Radiotherapy — Twice-daily thoracic radiotherapy at a dose of 54 Gy in 30 fractions with IMRT and VMAT
  Arms: Addition of thoracic consolidation radiotherapy to the maintenance therapy with PD-L1 inhibitor
Drug: atezolizumab or durvalumab — atezolizumab 1200 mg Q3W or durvalumab 1500 mg Q4W

SUMMARY:
This study is expected to enroll 182 patients with partial response or stable disease after first-line immunochemotherapy for extensive-stage small cell lung cancer and eligible for thoracic consolidation radiotherapy within 2 years. Patients were randomized 2:1 to immune single-agent maintenance therapy in combination with hyperfractionated high-dose radiotherapy and immune single-agent maintenance therapy after being assessed by the investigator as otherwise eligible for enrollment. Patients in both arms received maintenance therapy with the PD-L1 inhibitor, atezolizumab or dulvedolizumab, until disease progression, unacceptable toxicity, or loss of clinical benefit. Patients in the combined radiotherapy arm required hyperfractionated high-dose (54 Gy) radiotherapy twice daily for residual disease in the chest. Each patient will be followed for approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed written consent.
2. Age ≥ 18 years.
3. Confirmed Extensive Stage Small Cell Lung Cancer (ES-SCLC).
4. ECOG PS 0-1.
5. No previous systemic therapy except for induction immunochemotherapy for ES-SCLC.
6. Partial response or stable disease after 4-6 cycles of induction immunochemotherapy (PD-L1 inhibitor + cisplatin/carboplatin + etoposide). No more than 28 days between last tumor assessment before randomization and randomization.
7. Eligible for thoracic radiotherapy as assessed by the radiotherapy physician (The dose limits predicted for the organs at risk are as follows: bilateral lung V20 ≤ 25%, V5 ≤ 48%).
8. Patients with stable, asymptomatic CNS metastases are allowed.
9. Adequate bone marrow, renal function, and hepatic function.
10. Male or female patients of childbearing potential volunteered to use effective contraception during the study and within 6 months of the last dose of study drug.

Exclusion Criteria:

1. Prior thoracic radiotherapy.
2. History of interstitial lung disease (including but not limited to idiopathic pulmonary fibrosis), pneumonitis, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
3. Positive testing for hepatitis B virus surface antigen (HBV sAg), hepatitis C virus ribonucleic acid (HCV RNA), or human immunodeficiency virus (HIV).
4. Leptomeningeal metastasis.
5. Uncontrolled tumor-related pain.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
7. Malignancies other than NSCLC within 5 years prior to enrollment, with the exception of those treated with expected curative outcome.
8. Active or history of autoimmune disease or immune deficiency.
9. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to enrollment, unstable arrhythmias, or unstable angina.
10. Major surgical procedure other than for diagnosis within 4 weeks prior to enrollment or anticipation of need for a major surgical procedure during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2028-12-16 (Estimated); Study Completion 2028-12-16 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to the date of death due to any cause, assessed up to 4 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization to any documented progression or death due to any cause, whichever occurs first, assessed up to 4 years
Landmark analyses of survival | 1-year and 2-year landmark analysis of OS and 6-month and 1-year landmark analysis of PFS
Best overall response (BOR) | Up to 4 years
  BOR is the percentage of participants who have a CR or a PR, as determined by investigators according to RECIST v1.1.
Confirmed objective response rate (cORR) | Up to 4 years
  cORR is defined as either a confirmed CR or PR on two consecutive evaluations ≥ 4 weeks apart, as determined by investigators according to RECIST v1.1.
Incidence and severity of adverse events | From randomization to 30 days after the end of study treatment

IPD SHARING:
Plan to Share IPD: Yes
IPD related to article disclosure data
Supporting Information: Study Protocol
Time Frame: Available after publication
Access Criteria: Request by email to PI